CLINICAL TRIAL: NCT05378633
Title: The CyberChallenge Trial How Much is Too Much - What is the Role of Cyberknife Radiosurgery in Patients With Multiple Brain Metastases?
Acronym: CyberChallenge
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Head of Department, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The CyberChallenge Trial
Record Dates: First submitted 2022-01-24; First posted 2022-05-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Brain Metastases; Nsclc
Keywords: Metastases; Cyberknife; Lung Cancer
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment Arm (Experimental): Best Supportive Care + Stereotactic Radiotherapy of all Brain Metastases
  Interventions: Radiation: SRS
- Standard Treatment Arm (Other): Best Supportive Care ± Whole Brain Radiotherapy
  Interventions: Radiation: Whole Brain Radiotherapy

INTERVENTIONS:
Radiation: SRS — Stereotactic Radiotherapy (SRS)
  Arms: Experimental Treatment Arm
Radiation: Whole Brain Radiotherapy — Whole Brain Radiotherapy (WBRT)
  Arms: Standard Treatment Arm

SUMMARY:
Patients suffering from malignancies in advanced stages often develop brain metastases, which limit both the life span and the quality of life.

Therapy options for multiple brain metastases may vary and range from stereotactic radiosurgery (SRS), whole-brain radiotherapy (WBRT), chemotherapy, immunotherapy to palliative best supportive care. Especially the efficacy and toxicity of SRS compared to WBRT in patients with extensive brain metastases (>4) is not yet clear but of incremental relevance in this seriously ill cohort with a limited life span. These health-impaired patients might especially profit from a less toxic treatment that is also time sparing with 1 or few sessions in SRS versus 10 sessions in WBRT. On the other hand, no compromises in efficacy want to be done.

DETAILED DESCRIPTION:
In the present multicenter study, the benefit of SRS compared to conventional whole brain radiotherapy, each combined with best supportive care or best supportive care only, in patients with 4-15 brain metastases is to be prospectively investigated. The effect will be measured using quality-adjusted life-years (QUALY). Quality of life and overall survival are therefore primary endpoints. Secondary endpoints are the ability to perform basic activities of daily life (Barthel (ADL) index), progression-free survival, local and locoregional progression-free survival, extracranial progression, toxicity and its treatment, the recording of postherapeutic radiation-induced brain lesions (RIBL), long-term cognitive function, a possible salvage therapy as well as death from brain metastases. Furthermore, die CyberChallenge trial is linked to a translational program via BUB2 study. The BUB2 study conducts biobanking of blood, urine and resection or biopsy material, if available, as well as collects imaging material. This is to find diagnostic and prognostic biomarkers in our cancer patients via analyzing genetic, epigenetic and protein expression patterns as well as radiomics and correlating them to clinical data and therefore further push individualized patient care in brain metastases forward.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed malignant illness
* 4-15 suspect intracranial lesions, taking into consideration all available MRI series
* age ≥ 18 years of age
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Refusal of the patients to take part in the study
* Inability to tolerate irradiation consistent with the protocol
* Small-cell lung cancer (SCLC) or lymphoma as primary malignant illness
* >15 suspect intracranial lesions, taking into consideration all available MRI series
* leptomeningeal disease
* Previous radiotherapy of the brain
* Patients who have not yet recovered from acute high-grade toxicities of prior therapies
* Pregnant or lactating women
* Participation in another competing clinical study or observation period of competing trials, respectively
* MRI contraindication (i.e. cardiac pacemaker, implanted defibrillator, certain cardiac valve replacements, certain metal implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2025-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
overall survival | time from randomisation until the date of death from any cause, assesd up to 24 month
  number of alive patients
quality of life according to QLQ-C15 (questionaire for patients with advanced cancer referred for palliative radiotherapy | time from randomisation until the date of death from any cause, assesd up to 24 month
  changes in QLQ-C15 scores, scale is 1-100 points, 100 points representing maximum score
quality of life according to BN-20 (questionaire for patients with brain neoplasm) | time from randomisation until the date of death from any cause, assesd up to 24 month
  changes in BN-20 scores, scale is 1-100 points, 100 points representing maximum score

SECONDARY OUTCOMES:
functional independence assessed by the Barthel ADL index | time from randomisation until the date of death from any cause, assesd up to 24 month
  Changes in Barthel ADL index scores, scale 0-100 points
long-term cognitive Status (Hopkins Verbal Learning Test HVLT) | time from randomisation until the date of death from any cause, assesd up to 24 month
  Changes in HVLT scores (minimum 0, maximum 12)
development of radiation-induced brain lesions | time from randomisation until the date of death from any cause, assesd up to 24 month
  changes in amounts of Radiation-induced brain lesions
Radiation induced sideeffects | time from randomisation until the date of death from any cause, assesd up to 24 month
  changes in toxicity rates according to CTCAE 5.0
Overall survival | time from randomisation until the date of death from any cause, assesd up to 24 month
  amount of alive randomized patients enrolled in the trial
local progression of treated metastases | time from randomisation until the date of death from any cause, assesd up to 24 month
  detectable progressive disease of treated metastases
intracranial progression of leptomeningeal disease | time from randomisation until the date of death from any cause, assesd up to 24 month
  occurrence of leptomeningeal disease
intracranial progression of treated BM disease | time from randomisation until the date of death from any cause, assesd up to 24 month
  recurrence of treated BM disease
intracranial progression of new BM disease | time from randomisation until the date of death from any cause, assesd up to 24 month
  occurrence of new BM disease
Brain salvage during follow-up | time from randomisation until the date of death from any cause, assesd up to 24 month
  medical idication for whole brain Radiation after inital stereotactic radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, Prof., Principal Investigator — Head of Department
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No